CLINICAL TRIAL: NCT00579553
Title: Comparing Intramuscular Versus Vaginal Progesterone for Prevention of Preterm Birth.
Brief Title: Comparing IM vs. Vaginal Progesterone for Pre-term Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Progesterone75,643
Record Dates: First submitted 2007-12-18; First posted 2007-12-24 (Estimated); Results first posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Infant, Premature; Premature Birth
Keywords: Pre Term; Pre Term Birth; Premature Birth; Premature baby; High risk pregnancy; Progesterone; IM Progesterone; Vaginal Progesterone
MeSH Terms: conditions — Premature Birth | interventions — 17 alpha-Hydroxyprogesterone Caproate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intramuscular Progesterone (Active Comparator): Intramuscular Progesterone
  Interventions: Drug: Intramuscular Progesterone
- Vaginal Progesterone (Experimental): Vaginal Progesterone
  Interventions: Drug: Vaginal Progesterone

INTERVENTIONS:
Drug: Intramuscular Progesterone — Intramuscular Progestone: 17 alpha hydroxyprogesterone caproate: weekly 1 cc injections containing 250 mg of 17P
  Other Names: 17 alpha hydroxyprogesterone caproate
  Arms: Intramuscular Progesterone
Drug: Vaginal Progesterone — Vaginal Progesterone: 100 mg vaginal suppository daily
  Arms: Vaginal Progesterone

SUMMARY:
This is a randomized controlled trial comparing weekly intramuscular injection of 17 alpha hydroxylprogesterone caproate with daily vaginal progesterone in women with singleton pregnancies and history of prior spontaneous preterm birth in terms of maternal, fetal and neonatal outcomes.

Our aim is to assess the effects on maternal, fetal and neonatal outcomes of antenatal progesterone administered intramuscularly versus vaginally in women with singleton pregnancy and a history of prior preterm birth.

DETAILED DESCRIPTION:
This study is intended as a randomized controlled trial. Women with singleton pregnancies between 16 and 20 weeks 6 day will be randomized to one of two treatment groups.

Those randomized to weekly intramuscular progesterone will receive 250 mg of 17 alpha hydroxyprogesterone caproate every week in the clinic between randomization and delivery for those delivery preterm or 36 weeks 6 days.

While those randomized to vaginal progesterone will receive 100 mg vaginal progesterone daily at home. Vaginal progesterone to last between clinic visits will be provided to subject. Those women in the vaginal progesterone group will also be informed on how to obtain additional medication in case of missed clinic appointment. Treatment will be continued until 36 weeks 6 days or as dictated by date of preterm delivery.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies
* History of spontaneous preterm brith (between 20 weeks and 36 weeks 6 days)
* Gestational age between 16 weeks 0 days and 20 weeks 6 days.
* Signed consent to participate in the trial

Exclusion Criteria:

* Multiple Gestation
* Prior elective fetal reduction or planned termination
* Known spontaneous reduction to singleton
* Major fetal anomaly or known fetal chromosomal abnormalities
* Progesteone used this pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 174 (Actual)
Dates: Start 2006-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Elimian, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Derived] Elimian A, Smith K, Williams M, Knudtson E, Goodman JR, Escobedo MB. A randomized controlled trial of intramuscular versus vaginal progesterone for the prevention of recurrent preterm birth. Int J Gynaecol Obstet. 2016 Aug;134(2):169-72. doi: 10.1016/j.ijgo.2016.01.010. Epub 2016 Apr 18. PMID 27168167

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intramuscular Progesterone | Vaginal Progesterone
Started | 82 | 92
Completed | 66 | 79
Not Completed | 16 | 13
Not completed — Lost to Follow-up | 16 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intramuscular Progesterone | Vaginal Progesterone | Total
Number analyzed (Participants) | 66 | 79 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.6 (4.3) | 26.8 (4.7) | 26.3 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 79 | 145
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 66 | 79 | 145
Educational Level [Count of Participants; unit: Participants]
  College | 6 | 9 | 15
  High School | 38 | 44 | 82
  Less than high school | 22 | 26 | 48
Tobacco use [Count of Participants; unit: Participants]
  Tobacco use | 11 | 16 | 27
  No tobacco use | 55 | 63 | 118

OUTCOME MEASURES:

1. Primary Outcome: Preterm Birth
Description: Delivery before 37 weeks gestation.
Time Frame: From 16-20 weeks gestation through preterm delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Intramuscular Progesterone | Vaginal Progesterone
Number analyzed (Participants) | 66 | 79
Participants | 29 | 30

2. Secondary Outcome: Preterm Birth
Description: Delivery below 34 weeks gestation
Time Frame: From 16-20 weeks gestation through preterm delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Intramuscular Progesterone | Vaginal Progesterone
Number analyzed (Participants) | 66 | 79
Participants
  Delivery less than 34 weeks | 13 | 14
  Delivery less than 28 weeks | 7 | 8

3. Secondary Outcome: Gestational Age at Delivery
Description: Mean gestational age at delivery
Time Frame: From 16-20 weeks gestation through preterm delivery
Measure: Mean (Standard Deviation); unit: Weeks gestation
Arm/Group | Intramuscular Progesterone | Vaginal Progesterone
Number analyzed (Participants) | 66 | 79
Weeks gestation | 35.8 (4.7) | 36.3 (5.7)

4. Secondary Outcome: Mean Neonatal Birth Weight
Time Frame: At delivery
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Intramuscular Progesterone | Vaginal Progesterone
Number analyzed (Participants) | 66 | 79
grams | 2680.6 (840) | 2771.6 (1131)

ADVERSE EVENTS:
Arm/Group | Intramuscular Progesterone | Vaginal Progesterone
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/79
Other Adverse Events (participants affected / at risk) | 0/66 | 0/79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes